CLINICAL TRIAL: NCT01716767
Title: Acute Effect of Topical Menthol on Pain Symptoms in Slaughterhouse Workers With Symptoms of Carpal Tunnel Syndrome: Randomized Controlled Trial
Brief Title: Acute Effect of Topical Menthol on Carpal Tunnel Syndrome
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Principal Investigator, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRMA07
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; hand pain; wrist pain; arm pain; topical menthol
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Menthol; Analgesics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menthol (Experimental): Biofreeze topical gel containing 3.5% menthol
  Interventions: Other: Menthol
- Placebo (Placebo Comparator): Topical gel containing a menthol scent, but no active menthol
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Menthol — The gel will be applied at 2.5 ml per 500 cm2 to the hand, wrist and forearm
  Other Names: Topical analgesic
  Arms: Menthol
Other: Placebo — The gel will be applied at 2.5 ml per 500 cm2 to the hand, wrist and forearm
  Arms: Placebo

SUMMARY:
Topical menthol gels are classified 'topical analgesics' and are used to relieve pain of the musculoskeletal system. However, double-blind randomized controlled trials are lacking. Here the investigators examine - in a double-blind randomized controlled cross-over trial - the acute effect of topical menthol (Biofreeze) and placebo (gel with a menthol scent) on pain symptoms in slaughterhouse workers with symptoms of Carpal Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* positive Phalen test
* positive Tinel test
* nocturnal hand/wrist pain
* pain intensity of at least 4 in the hand/wrist
* the pain should have lasted at least 3 months

Exclusion Criteria:

* pregnancy
* life-threatening disease

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in arm/hand pain intensity (scale 0-10) during work | change from before to after (average of 1,2 and 3 hours after) application of the gel
  the participant rates "pain intensity during the last hour" on a scale from 0-10 immediately before, and 1,2,3 hours after application of the gel. The primary outcome is the change from before to after (average of 1,2 and 3 hours after) application of the gel

SECONDARY OUTCOMES:
GROC | 3 hours after application of the gel
  Global Rating of Change (GROC) on a scale from - 5(much worsening of pain) to 5(much improvement of pain)

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — Professor
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark